CLINICAL TRIAL: NCT02577432
Title: Two Syringe Spinal Anesthesia Technique for Cesarean Section: A Controlled Randomized Study of a Simple Way to Achieve More Satisfactory Block and Less Hypotension
Brief Title: Two Syringe Spinal Anesthesia Technique for Cesarean Section: A Simple Way to Achieve More Satisfactory Block and Less Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soliman Fakeeh Hospital (Other)
Responsible Party: Principal Investigator, Dr. Amr Aly Ismail Keera, Assistant professor, Dr. Soliman Fakeeh Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01/REC/2013
Record Dates: First submitted 2015-10-10; First posted 2015-10-16 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Cesarean Section
Keywords: spinal anesthesia
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (S) separate. (Active Comparator): fentanyl and hyperbaric bupivacaine (sequentially)
  Interventions: Drug: fentanyl; Drug: Hyperbaric bupivacaine
- (M) mixed (Active Comparator): fentanyl and hyperbaric bupivacaine.(mixed)
  Interventions: Drug: fentanyl; Drug: hyperbaric bupivacaine

INTERVENTIONS:
Drug: fentanyl — Give 25 micro grams fentanyl intrathecal with one syringe. Then immediately give 10 mg hyperbaric bupivacaine intrathecally with an other syringe.
  Arms: (S) separate.
Drug: fentanyl — Mix 25 micro grams fentanyl with 10 mg hyperbaric bupivacaine in one syringe. Give them intrathecally.
  Arms: (M) mixed
Drug: Hyperbaric bupivacaine — Give 25 micro grams fentanyl intrathecal with one syringe. Then immediately give 10 mg hyperbaric bupivacaine intrathecally with an other syringe.
  Arms: (S) separate.
Drug: hyperbaric bupivacaine — Mix 25 micro grams fentanyl with 10 mg hyperbaric bupivacaine in one syringe. Give them intrathecally.
  Arms: (M) mixed

SUMMARY:
Background: Poor spinal anaesthesia block is common and is difficult to manage; so a technique to minimize its incidence is advisable. Hypotension is the commonest problem with spinal anesthesia. Multiple trials to prevent or combat hypotension using positional changes, fluid therapy and the use of vasopressors were tried. However, the drug choice and mode of administration as either bolus or infusion is still a matter of debate.

Objectives: To compare the outcome of spinal injection of hyperbaric bupivacaine and fentanyl separately to standard injection of mixed fentanyl with hyperbaric bupivacaine.

Design: A randomized, controlled clinical trial.

Setting: Single medical center from 5/2013 to 10/2014.

Patients & Methods: 124 parturient scheduled for elective cesarean section (CS) were randomly allocated into two groups, each 62 parturient: Group M received spinal anesthesia using 10 mg bupivacaine 0.5% premixed with 25 µg fentanyl in the same syringe and Group S received 25 µg fentanyl in one syringe and 10 mg bupivacaine 0.5% without barbotage in a second syringe. Intravenous fluid co-load with 15 ml/kg warm lactated ringer solution was started as fast drip during, and continued after spinal anesthesia.

Patients were monitored for hemodynamic parameters, time of sensory onset and height of maximum sensory block, lower limb motor blockade was scored using modified Bromage scale and the frequency of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Parturient at full term.
* Must be elective cesarean section.
* Must be uncomplicated pregnancy

Exclusion Criteria:

* Body weight <50 kg or >90 kg
* Height ˂150 cm or >170 cm.
* Pre-eclampsia.
* Any major systemic disease.
* Contraindication to regional anesthesia.
* Allergy to used medications.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of parturients needed more analgesics (unsatisfactory block) using Ochsner Health System. | intraoperative
incidence of hypotension | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Keera, MD, Principal Investigator — Dr. Benha Faculty of Medicine